CLINICAL TRIAL: NCT02620709
Title: The KaHOLO Project: Preventing Cardiovascular Disease in Native Hawaiians
Acronym: KaHOLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Hawaii (Other)
Collaborators: I Ola Lahui, Inc. (Other); Ke Ola Mamo (Other); University of Washington (Other); Hui No Ke Ola Pono, Inc. (Other); Kula No Na Po'e Hawaii (Other)
Responsible Party: Principal Investigator, Joseph Keawe'aimoku Kaholokula, Chair and Associate Professor, University of Hawaii
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KaHOLO Project
Record Dates: First submitted 2015-11-23; First posted 2015-12-03 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: Native Hawaiians; Community-based participatory research; Health disparities; Minority populations; Chronic disease
MeSH Terms: conditions — Hypertension; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hula intervention (Experimental): Participants randomized to the intervention arm will receive the 6-month KaHOLO Program within 1 week of baseline data collection. The first 3 months of the KaHOLO was designed and standardized as a culturally-based PA, which includes 12 weeks of hula lessons. These hula lessons consist of two 60 minute classes per week over 12 weeks. Each hula lesson will consist of 15 participants, providing with the opportunity to engage in social support network.
  The last three months of the program will be reduced to once a week sessions. One week will consist of hula lessons for 60 minutes. The remaining 3 weeks will consist of the intervention group meeting for 45 minutes with the community-peer educator.
  Interventions: Behavioral: Hula intervention
- Wait-List Control (No Intervention): After baseline data collection and education, participants randomized to the wait-list control arm will not receive the KaHOLO Program while their counterparts who were randomized to the intervention arm are undergoing the intervention program. Thus, they will not receive the intervention for 6 months until after the intervention arm is completed and their 6 month follow-up data collection is completed. They will not receive any other intervention from us during the 6 month period but they will be instructed to continue with their routine medical care as usual.

INTERVENTIONS:
Behavioral: Hula intervention — Hula and heart health education
  Arms: Hula intervention

SUMMARY:
This project is a community-engaged, randomized control trial of hula, the indigenous dance form of Native Hawaiians (NH), among 250 NHs with hypertension living in Hawaii and Washington State. Investigators will compare the effects of a 6-month intervention, called the KaHOLO Program, delivered by trained peer educators to a wait-list control condition on blood pressure and 10-year cardiovascular risk. The intervention will be comprised of hula plus hypertension self-care education program. Investigators will also examine the mediating effects of health behaviors, self-regulation, psychosocial, and socio-cultural factors on blood pressure reduction. The ultimate goal is to develop and test a culturally-appropriate, acceptable, and effective intervention that can be delivered and sustained in community settings.

DETAILED DESCRIPTION:
Native Hawaiians (NH) have higher rates of chronic diseases, such as cardiovascular disease (CVD), diabetes, and cancer. Hypertension (HTN), an important modifiable risk factor for CVD, is 70% higher in Native Hawaiians (NH) than in Whites. In fact, NH are 3-4 times more likely to develop CVD conditions, such as stroke and coronary heart disease, and at a younger age. In addition to prescribed medication, improvements in HTN can be achieved through increased physical activity (PA) and self-management education (e.g. stress management, reduces sodium intake, weight-loss, and smoking cessation). Yet, many commonly prescribed PA, such as jogging and use of treadmills, are difficult for NH to initiate and maintain because of socioeconomic barriers and lack of alignment with NH preferred modes of living and cultural values (i.e. familial interdependence, group-based PA, cultural PA).

This research study uses hula, the traditional dance form of NH and hallmark of NH culture, as the PA basis for a culturally relevant and sustainable CVD prevention program targeting HTN management. Hula training is popular, not only Hawai'i, but across the U.S. through the 784 hālau hula (hula schools) found in most States. Using a community-based participatory research (CBPR) framework, a hula-based CVD health intervention was strongly endorsed by Kumu hula (hula experts and guardians of hula traditions), NH individuals, and communities. Further, hula was determined to yield metabolic equivalent of energy expenditure as a moderate and vigorous intensity PA. Data from a pilot CBPR randomized control trial (RCT) study found that 60 minutes of hula training twice a week for 12 weeks reduced systolic blood pressure (BP) by 7.5 mmHg (SD=16.5) more than the control group, but the long-term effects were mixed and the study did not assess CVD risk.

Interestingly, the pilot intervention also improved social functioning, reduced physical pain, and perceived racial discrimination, suggesting a possible psychosocial and socio-cultural mechanism by which the intervention affects BP. In this study a CBPR guided RCT of 250 NH with physician-diagnosed HTN in Hawai'i and Washington State is offered. The effects will be compared of a 6-month intervention that combines hula training and brief culturally-tailored HTN self-management education delivered by peer educators and Kumu hula to a wait-list control group in reducing systolic BP and CVD risk scores. It will also be determined the mediating effects of health behaviors (e.g., smoking), self-regulation, and psychosocial (e.g., social support), and socio-cultural factors (e.g., perceived racism) on blood pressure reduction. The goal is to build on the existing widespread infrastructure of hālau hula and NH organizations to deliver a sustainable, culturally-preferred CVD prevention program.

ELIGIBILITY:
Inclusion Criteria:

* Native Hawaiian ancestry
* Physician diagnosed HTN
* Continued SBP>140
* Physicians approval to participate in moderate PA
* No prior CVD history

Exclusion Criteria:

* Pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in participants' systolic blood pressure at each time frame from baseline | 3 months, 6 months, and 12 months

SECONDARY OUTCOMES:
Change in participants' Framingham Risk Score of 10 year CVD risk at each time frame from baseline | 3 months, 6 months, and 12 months

OTHER OUTCOMES:
Number of Participants with decreased scores on the Perceived Ethnic Discrimination Scale | 3 months, 6 months, and 12 months
Number of Participants with improved monthly physical activity levels as assessed by the Physical Activity Questionnaire | 3 months, 6 months, and 12 months
Number of participants with increased scores on the Medical Outcomes Study (MOS) 36-item Social Support Survey | 3 months, 6 months, and 12 months
Number of participants with decreased scores on the Perceived Stress Scale | 3 months, 6 months, and 12 months
Number of participants with increased scores of the Exercise Self-Efficacy Scale | 3 months, 6 months, and 12 months
Number of participants with increased scores on the Native Hawaiian Identity Scale | 3 months, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Kaholokula, PhD, Principal Investigator — University of Hawaii
Locations (1):
- University of Hawaii, John A Burns School of Medicine, Department of Native Hawaiian Health, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Railey AF, Muller C, Noonan C, Schmitter-Edgecombe M, Sinclair K, Kim C, Look M, Kaholokula JK. Cost Effectiveness of a Cultural Physical Activity Intervention to Reduce Blood Pressure Among Native Hawaiians with Hypertension. Pharmacoecon Open. 2022 Jan;6(1):85-94. doi: 10.1007/s41669-021-00291-6. Epub 2021 Aug 13. PMID 34389923
- [Derived] Kaholokula JK, Look MA, Wills TA, de Silva M, Mabellos T, Seto TB, Ahn HJ, Sinclair KA, Buchwald D; Ka-HOLO Project. Ka-HOLO Project: a protocol for a randomized controlled trial of a native cultural dance program for cardiovascular disease prevention in Native Hawaiians. BMC Public Health. 2017 Apr 17;17(1):321. doi: 10.1186/s12889-017-4246-3. PMID 28415975